CLINICAL TRIAL: NCT02546375
Title: A RETROSPECTIVE OBSERVATIONAL RESEARCH STUDY TO DESCRIBE THE REAL WORLD USE OF BOSUTINIB IN THE UK AND NETHERLANDS
Brief Title: A Study To Describe The Real World Use Of Bosutinib In The UK And Netherlands
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: pH Associates (Unknown)
Responsible Party: Sponsor
Other Study IDs: B1871052
Record Dates: First submitted 2015-08-26; First posted 2015-09-10 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Chronic Myeloid Leukaemia
Keywords: Bosutinib; chronic myeloid leukaemia; retrospective; observational
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Myeloid Leukaemia: Patients diagnosed with chronic myeloid leukaemia treated with Bosutinib
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib — Bosutinib 100mg film-coated tablets; Bosutinib 500mg film-coated tablets Dosage as prescribed at treating institution; (observational study)
  Other Names: Bosulif

SUMMARY:
The purpose of this study is to describe the efficacy and safety of bosutinib in patients with chronic myeloid leukaemia used in a real world setting

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ph+ CML aged ≥18 years at bosutinib initiation.
* Prescribed bosutinib (irrespective of the phase of their disease) EITHER in normal clinical practice since it received marketing authorisation (27th March 2013) by the EMA11 OR via the compassionate use programme prior to marketing authorization.
* Where required, evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Prescribed bosutinib as part of an interventional clinical trial programme.
* Initiated on bosutinib less than 3 months prior to data collection taking place.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CML out-patient clinics
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United Kingdom (3):
  - Royal Liverpool Hospital, Liverpool, Merseyside
  - Hammersmith Hospital, London
  - Nottingham University Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1871052&StudyName=A%20Retrospective%20Observational%20Research%20Study%20To%20Describe%20The%20Real%20World%20Use%20Of%20Bosutinib%20In%20The%20Uk%20And%20Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Bosutinib: Participants with Philadelphia chromosome-positive chronic myeloid leukemia (CML) receiving imatinib, dasatinib or nilotinib prior to enrollment in the study, who were treated with single daily oral dose of Bosutinib 100 to 500 milligram (mg), were observed up to a maximum duration of 5.5 years. Dosage and use of Bosutinib was based on treating physician, according to approved Summary of Product Characteristics (SmPC).
Period: Overall Study
Arm/Group | Bosutinib
Started | 87
Completed | 87
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants with Philadephia chromosome positive CML in chronic phase received at least 1 dose of Bosutinib.
Groups:
- Bosutinib: Participants with Philadelphia chromosome-positive CML receiving imatinib, dasatinib or nilotinib prior to enrollment in the study, who were treated with single daily oral dose of Bosutinib 100 to 500 mg, were observed up to a maximum duration of 5.5 years. Dosage and use of Bosutinib was based on treating physician, according to approved SmPC.
Arm/Group | Bosutinib
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (14.3) [24.8 to 90.1]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 40
  Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Cumulative Complete Haematological Response (CHR)
Description: Haematological response used blood sample of the participants to evaluate response to treatment for CML. Based on the European LeukemiaNet (ELN) 2013 definition: CHR is defined as platelet count less than (<) 450*10^9 per liter, white blood cells count <10*10^9 per liter, no immature granulocytes and <5 percent (%) basophils on differential and a non-palpable spleen.
Time Frame: Baseline up to 5.5 years
Population: All enrolled participants with Philadephia chromosome positive CML in chronic phase received at least 1 dose of Bosutinib. Here, number of participants analyzed (N) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 84
percentage of participants | 93

2. Primary Outcome: Percentage of Participants With Cumulative Partial Haematological Response (PHR)
Description: Haematological response used blood sample of the participants to evaluate response to treatment for CML.
Time Frame: Baseline up to 5.5 years
Population: All enrolled participants with Philadephia chromosome positive CML in chronic phase received at least 1 dose of Bosutinib. Here, N signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 84
percentage of participants | 94

3. Primary Outcome: Percentage of Participants With Cumulative Complete Cytogenetic Response (CCyR)
Description: Cytogenetic response (CyR) used bone marrow/blood sample of the participants to evaluate response to treatment for CML. Based on the ELN 2013 definition: CyR was measured by chromosome banding analysis (CBA) or fluorescence in situ hybridisation (FISH). CCyR was indicated by absence of Philadelphia chromosome positive (Ph+) cells metaphases from FISH of blood interphase cell nuclei.
Time Frame: Baseline up to 5.5 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 84
percentage of participants | 67

4. Primary Outcome: Percentage of Participants With Cumulative Minor Cytogenetic Response (MCyR)
Description: CyR used bone marrow/blood sample of the participants to evaluate response to treatment for CML. Based on the ELN 2013 definition: CyR was measured by CBA or FISH. MCyR was indicated by presence of 36-65% Ph+ cells from CBA of bone marrow metaphases.
Time Frame: Baseline up to 5.5 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 84
percentage of participants | 77

5. Primary Outcome: Percentage of Participants With Cumulative Minimal Cytogenetic Response (mCyR)
Description: CyR used bone marrow/blood sample of the participants to evaluate response to treatment for CML. Based on the ELN 2013 definition: CyR was measured by CBA or FISH. mCyR was indicated by presence of 66-95% Ph+ cells from CBA of bone marrow metaphases.
Time Frame: Baseline up to 5.5 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 84
percentage of participants | 80

6. Primary Outcome: Percentage of Participants With Cumulative Partial Cytogenetic Response (PCyR)
Description: CyR used bone marrow/blood sample of the participants to evaluate response to treatment for CML. Based on the ELN 2013 definition: CyR was measured by CBA or FISH. PCyR was indicated by presence of 1-35% Ph+ cells from CBA of bone marrow metaphases.
Time Frame: Baseline up to 5.5 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 84
percentage of participants | 77

7. Primary Outcome: Percentage of Participants With Cumulative Complete Molecular Response 4.0 (MR4.0)
Description: Molecular response used blood sample of the participants to evaluate response to treatment for CML. Based on the ELN 2013 definition: Molecular response used breakpoint cluster region/Abelson (BCR-ABL1) transcript measured by real time quantitative polymerase chain reaction (RT-Q-PCR). Evaluation was expressed as percentage of ratio of BCR-ABL1 transcripts to ABL1 transcripts according to the international scale (IS) or the ratio of BCR/ABL1 transcripts to other internationally recognized control transcripts levels. MR4.0 was defined and recorded as detectable disease with <0.01% BCR-ABL1 transcripts on IS or undetectable disease in cDNA with greater than (>) 10,000 ABL1 transcripts in the same volume of cDNA used to test for BCR-ABL1 transcripts.
Time Frame: Baseline up to 5.5 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 84
percentage of participants | 33

8. Primary Outcome: Percentage of Participants With Cumulative Complete Molecular Response 4.5 (MR4.5)
Description: Molecular response used blood sample of the participants to evaluate response to treatment for CML. Based on the ELN 2013 definition: Molecular response used breakpoint cluster region/Abelson (BCR-ABL1) transcript measured by real time quantitative polymerase chain reaction (RT-Q-PCR). Evaluation was expressed as percentage of ratio of BCR-ABL1 transcripts to ABL1 transcripts according to the international scale (IS) or the ratio of BCR/ABL1 transcripts to other internationally recognized control transcripts levels. MR4.5 was defined and recorded as detectable disease with <0.0032% BCR-ABL1 transcripts on IS or undetectable disease in cDNA with >32,000 ABL1 transcripts in the same volume of cDNA used to test for BCR-ABL1 transcripts.
Time Frame: Baseline up to 5.5 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 84
percentage of participants | 27

9. Primary Outcome: Percentage of Participants With Cumulative Major Molecular Response (MMR)/Molecular Response 3.0 (MR3.0)
Description: Molecular response used blood sample of the participants to evaluate response to treatment for CML. Based on the ELN 2013 definition: Molecular response used breakpoint cluster region/Abelson (BCR-ABL1) transcript measured by real time quantitative polymerase chain reaction (RT-Q-PCR). Evaluation was expressed as percentage of ratio of BCR-ABL1 transcripts to ABL1 transcripts according to the international scale (IS) or the ratio of BCR/ABL1 transcripts to other internationally recognized control transcripts levels. MMR was defined as a BCR-ABL1 to ABL1 less than or equal to (<=) 0.1% on the IS.
Time Frame: Baseline up to 5.5 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 84
percentage of participants | 55

10. Secondary Outcome: Percentage of Participants With Treatment Related Adverse Events (AEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to Bosutinib in a participant who received Bosutinib. Relatedness to Bosutinib was assessed by the investigator.
Time Frame: Baseline up to 5.5 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 87
percentage of participants | 94

11. Secondary Outcome: Percentage of Participants With Treatment Related Adverse Events (AEs) Greater Than or Equal to Grade 3
Description: Treatment-related AE was any untoward medical occurrence attributed to Bosutinib in a participant who received Bosutinib. AE was assessed according to maximum severity grading based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. Grade 1 =mild; Grade 2 =moderate; within normal limits, Grade 3 =severe or medically significant but not immediately life-threatening; Grade 4 =life-threatening or disabling; urgent intervention indicated; Grade 5 =death.
Time Frame: Baseline up to 5.5 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 87
percentage of participants | 21

12. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the duration between initiation of Bosutinib therapy and date of progression estimated by the treating physician or death of participant (all causes combined). Progression was defined as change from chronic phase of CML (CP-CML) to accelerated phase of CML (AP-CML) or to blast crisis of CML (BC-CML). CP-CML is frequently asymptomatic and diagnosed with <10% blasts. Based on the ELN 2013 definition: AP-CML was defined by the presence of blast cells between 15-29% or blast cells plus promyelocytes >30%, with blasts <30% in blood or bone marrow, platelet count <100*10^9 or clonal chromosome abnormalities in Ph+ cells. BC-CML was defined as blasts in blood or bone marrow >=30%, extramedullary blast proliferation (excluding spleen), large foci or clusters of blasts in bone marrow biopsy. Participants who were alive at the date of last assessment were censored on the date of data collection.
Time Frame: Year 1, 2, 3
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Bosutinib
Number analyzed (Participants) | 87
years | NA [NA to NA] — Median and 95% Confidence interval (C.I.) were not reached due to small number of events.

13. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from initiation of Bosutinib therapy to date of death (all causes combined). For participants who were alive or lost to follow-up (LTFU), overall survival was censored on the date of data collection or date LTFU, respectively.
Time Frame: From baseline up to 1 Year, baseline up to Year 2, baseline up to Year 3
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Bosutinib
Number analyzed (Participants) | 87
years | NA [NA to NA] — Median and 95% C.I. were not reached due to small number of events.

14. Secondary Outcome: Percentage of Participants With Disease Progression
Description: Progression was defined as change from CP-CML to AP-CML or to BC-CML. CP-CML is frequently asymptomatic and diagnosed with <10% blasts. Based on the ELN 2013 definition: AP-CML was defined by the presence of blast cells between 15-29% or blast cells plus promyelocytes >30%, with blasts <30% in blood or bone marrow, platelet count <100*10^9 or clonal chromosome abnormalities in Ph+ cells. BC-CML was defined as blasts in blood or bone marrow >=30%, extramedullary blast proliferation (excluding spleen), large foci or clusters of blasts in bone marrow biopsy.
Time Frame: Year 1, 2, 3
Population: All enrolled participants with Philadephia chromosome positive CML in chronic phase received at least 1 dose of Bosutinib. Here, N signifies those participants who were evaluable for this outcome measure and number analyzed (n) signifies those participants who were evaluable at specified time points only.
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 84
percentage of participants
  1 year: number analyzed (Participants) | 66
  1 year | 3
  2 year: number analyzed (Participants) | 36
  2 year | 3
  3 year: number analyzed (Participants) | 12
  3 year | 0

15. Secondary Outcome: Percentage of Participants With Permanent Discontinuation From Bosutinib Therapy
Time Frame: Baseline up to 5.5 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 87
percentage of participants
  Adverse event | 14
  Loss of response | 5
  Treatment failure | 11
  Participant request | 2
  Death | 2
  Disease progression | 1
  Other | 2

16. Secondary Outcome: Cross-Intolerance Between Bosutinib and Previous Therapy
Description: Cross-intolerance was defined as percentage of participants who permanently discontinued bosutinib due to an adverse event which also resulted in discontinuation of a previous treatment (imatinib, dasatinib, nilotinib).
Time Frame: Baseline up to 5.5 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 87
percentage of participants | 1.1

17. Secondary Outcome: Mean Dose of Bosutinib at Initiation of Treatment
Time Frame: Baseline up to 5.5 years
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: milligram per day
Arm/Group | Bosutinib
Number analyzed (Participants) | 87
milligram per day | 331.0 (126.6)

18. Secondary Outcome: Relative Bosutinib Dose Intensity
Description: Relative dose intensity was defined as the percentage of daily dose received over the expected daily dose of the study drug.
Time Frame: Baseline up to 5.5 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of daily dose
Arm/Group | Bosutinib
Number analyzed (Participants) | 87
percentage of daily dose | 66

19. Secondary Outcome: Duration of Bosutinib Therapy
Description: The duration from initiation of Bosutinib therapy up to the end of Bosutinib therapy was reported in this outcome measure.
Time Frame: Baseline up to 5.5 years
Population: as for baseline characteristics
Measure: Median (Full Range); unit: months
Arm/Group | Bosutinib
Number analyzed (Participants) | 87
months | 15.6 [0.3 to 66.0]

ADVERSE EVENTS:
Time Frame: Baseline up to 5.5 years
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Bosutinib
Serious Adverse Events (participants affected / at risk) | 17/87
Other Adverse Events (participants affected / at risk) | 81/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib (N=87)
Anaemia (Blood and lymphatic system disorders) | 0
Creatinine increased (Blood and lymphatic system disorders) | 0
Neutropenia (Blood and lymphatic system disorders) | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 0
Cardiac failure (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 0
Abdominal Distension (Gastrointestinal disorders) | 0
Abdominal pain (Gastrointestinal disorders) | 0
Constipation (Gastrointestinal disorders) | 0
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 0
Nausea (Gastrointestinal disorders) | 0
Vomiting (Gastrointestinal disorders) | 1
Alopecia (General disorders) | 0
Asthenia (General disorders) | 0
Chest pain (General disorders) | 1
Fatigue (General disorders) | 0
Oedema (General disorders) | 0
Pain (General disorders) | 0
Pyrexia (General disorders) | 0
Other (General disorders) | 1
Alanine aminotransferase increased (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 0
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0
Dizziness (Nervous system disorders) | 0
Headache (Nervous system disorders) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0
Rash (Skin and subcutaneous tissue disorders) | 0
Pregnancy (Reproductive system and breast disorders) | 1
Pyelonephritis (Renal and urinary disorders) | 1
Diseases of the eye (Eye disorders) | 1
Lack of efficacy (General disorders) | 4
Haematological - not determined (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib (N=87)
Anaemia (Blood and lymphatic system disorders) | 3
Creatinine increased (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Atrial fibrillation (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 0
Hypertension (Cardiac disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 45
Dyspepsia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 4
Alopecia (General disorders) | 3
Asthenia (General disorders) | 1
Chest pain (General disorders) | 7
Fatigue (General disorders) | 16
Oedema (General disorders) | 1
Pain (General disorders) | 5
Pyrexia (General disorders) | 1
Other (General disorders) | 0
Alanine aminotransferase increased (Hepatobiliary disorders) | 15
Hepatotoxicity (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 0
Respiratory tract infection (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 15
Lack of efficacy (General disorders) | 10
Haematological - not determined (General disorders) | 4
Depression (Nervous system disorders) | 2
Diseases of the eye (Eye disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 2
Altered skin sensation (Skin and subcutaneous tissue disorders) | 1
Breaking nails (Skin and subcutaneous tissue disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Exostosis - benign growths of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fever (General disorders) | 1
Flu like symptoms (Infections and infestations) | 1
Medication error (General disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Rigors associates with extreme tiredness and thirst (General disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Sleep disturbance (Nervous system disorders) | 1
(General disorders) | 1
Unusual taste in mouth (Gastrointestinal disorders) | 1
Vitamin D deficiency (Musculoskeletal and connective tissue disorders) | 1
Weight gain (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.